CLINICAL TRIAL: NCT02550938
Title: Primer Aligner Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-300307-00
Record Dates: First submitted 2015-07-23; First posted 2015-09-16 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- 7 Aligner Cohort weartime 1 (Experimental): Seven Aligner cohort will change aligners at a designated interval Invisalign is the intervention.
  Interventions: Device: Invisalign
- 7 Aligner Cohort weartime 2 (Experimental): Seven Aligner cohort will change aligners at a modified interval Invisalign is the intervention.
  Interventions: Device: Invisalign
- 12 aligner cohort weartime 1 (Experimental): Twelve Aligner cohort will change aligners at a designated interval Invisalign is the intervention.
  Interventions: Device: Invisalign
- 12 aligner cohort weartime 2 (Experimental): Twelve Aligner cohort will change aligners at a modified interval Invisalign is the intervention.
  Interventions: Device: Invisalign

INTERVENTIONS:
Device: Invisalign — The Invisalign® System consists of a series of clear plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. Each aligner is worn for a defined period of time , then replaced by the next in the series until the final position is achieved. For years, orthodontists and dentists have used removable appliances for orthodontic treatment. Today, with the application of computer technology and custom manufacturing, Invisalign treats a broader range of cases with greater precision.

SUMMARY:
To demonstrate that a primer aligner product can achieve similar results to the currently marketed product.

DETAILED DESCRIPTION:
The Invisalign® System consists of a series of clear plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. Each aligner is worn for about two weeks, then replaced by the next in the series until the final position is achieved. For years, orthodontists and dentists have used removable appliances for orthodontic treatment. Today, with the application of computer technology and custom manufacturing, Invisalign treats a broader range of cases with greater precision.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have fully erupted dentition
* Age range ≥18 years old (Adult subject)
* Subjects who are indicated for either: 5, 7, 10, or 12 aligner sets

Exclusion Criteria:

* Subject who has unerupted, erupting, partially erupted dentition (except for 2nd and 3rd molars)
* Subject who has mixed dentition
* Subject with periodontal disease
* Subject with active caries
* Subject with Temporomandibular Joint Disorders symptoms
* Subject has undergone pre-treatment with any orthodontic appliance 3 months prior to the start of treatment
* Subject has undergone any accelerated orthodontic treatment prior to or during treatment as part of this study
* Subject has known allergy to latex or plastic
* Subjects who are pregnant or will become pregnant during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-05; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Moneim, DDS, Principal Investigator — Los Gatos Dental Center
Locations (19):
- United States (13):
  - Wood Orthodontics, Anthem, Arizona
  - Cooke Orthodontics, Napa, California
  - The Orthodontic Center, Oakland, California
  - Green Dentistry, San Francisco, California
  - Align Technology, Inc., San Jose, California
  - Posner, Henderson & Goslee Dentistry, Bristol, Connecticut
  - Feldman Orthodontics, Cheshire, Connecticut
  - Comizio Orthodontics, Eastchester, New York
  - Magic Touch Orthodontist, Little Neck, New York
  - Meadowbrook Dental Care, Mineola, New York
  - Wenger Orthodontics, Mayfield Heights, Ohio
  - Dental One Reston, Reston, Virginia
  - DMG Dental Design, Bothell, Washington
- United Kingdom (6):
  - Anglia Orthdontics, Cambridge, England
  - Bluebell Dental Practice, Chigwell, England
  - Dream Smile Dental Clinic, London, England
  - High Street Dental Care, Melton Mowbray, Leicestershire
  - Brixworth Dental Practice, Brixworth, Northampton
  - Cherrybank Dental Spa, Edinburgh, Scotland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2
Started | 44 | 85 | 43 | 81
Completed | 36 | 78 | 31 | 70
Not Completed | 8 | 7 | 12 | 11
Not completed — Lost to Follow-up | 8 | 7 | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2 | Total
Number analyzed (Participants) | 36 | 78 | 31 | 70 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 78 | 30 | 66 | 209
  >=65 years | 1 | 0 | 1 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 55 | 27 | 45 | 154
  Male | 9 | 23 | 4 | 25 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 50 | 20 | 36 | 126
  United Kingdom | 16 | 28 | 11 | 34 | 89

OUTCOME MEASURES:

1. Primary Outcome: Total Treatment Time
Description: Total treatment time was measured in days. The less days a subject was in treatment, the better.
Time Frame: Approximately 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2
Number analyzed (Participants) | 36 | 78 | 31 | 70
days | 197.4167 (102.0774) | 225.7 (108.463) | 326.9355 (151.414) | 294.1111 (181.7863)

2. Primary Outcome: Rate of Refinement
Description: Rate of Refinement was how often subjects in each cohort required additional aligners in (in addition to their originally prescribed aligners) to treat the malocclusion. For example, if a subject was originally prescribed 20 aligners for treatment, but then needed 10 more aligners, the 10 extra aligners would be considered the "refinement." The Rate of Refinement for each cohort was measured as the total number of additional aligners required to complete orthodontic treatment divided by the total number of aligners that were initially prescribed to complete treatment, multiplied by 100. The smaller the rate of refinement (%), the better.
Time Frame: Approximately 1 year
Measure: Mean (Standard Deviation); unit: percentage of refinement
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2
Number analyzed (Participants) | 36 | 78 | 31 | 70
percentage of refinement | 0.25 (0.439155) | 0.263158 (0.446258) | 0.419355 (0.50161) | 0.527778 (0.506309)

3. Other Pre Specified Outcome: Subject Satisfaction.
Description: (Observational, not used in data analysis). Subjects filled out a Quality of Life Survey with a scale rating of 1 (very difficult) to 5 (very easy) on how easy the product was to use and their orthodontic experience to date. A higher score on the scale meant a better outcome.
Time Frame: Approximately 1 year
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2
Number analyzed (Participants) | 36 | 78 | 31 | 70
score on a scale | 3.499 (2.473797384) | 3.156 (3.409) | 4.632 (4.499) | 4.499 (3.499)

4. Other Pre Specified Outcome: Doctor Survey Results.
Description: (Observational, not used in data analysis). Doctors filled out a Doctor Survey with a scale rating of 1 (very difficult) to 5 (very easy) on how easy the product was to use and their satisfaction with the product. A higher score on the scale meant a better outcome.
Time Frame: Approximately 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2
Number analyzed (Participants) | 36 | 78 | 31 | 70
score on a scale | 3.139 (1.4702645) | 2.899 (1.330019318) | 3.139 (3.1760840) | 4.499 (1.7756956)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the entire duration each subjects' participation in the clinical study, from enrollment until completion, an average of 262 days.
Arm/Group | 7 Aligner Cohort Weartime 1 | 7 Aligner Cohort Weartime 2 | 12 Aligner Cohort Weartime 1 | 12 Aligner Cohort Weartime 2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/85 | 0/43 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/85 | 0/43 | 0/81
Other Adverse Events (participants affected / at risk) | 0/44 | 0/85 | 0/43 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT02550938/Prot_000.pdf